CLINICAL TRIAL: NCT02242084
Title: Thrombolysis in Ischemic Spinal Cord Stroke
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, israel Steiner, Head of Neurology Department, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK 23 - 14
Record Dates: First submitted 2014-09-14; First posted 2014-09-16 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Motor Weakness in Two or Four Limbs; Damage in the Anterior Spinal Artery (ASA); Temperature and Superficial Sensation; Urinary Retention or Bowel Disorder
MeSH Terms: conditions — Urinary Retention; Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Alteplase treatment (Experimental): All subject who enter the trial will receive treatment with Alteplase along with questionnaire.
  Interventions: Drug: Intravenuse Alteplase

INTERVENTIONS:
Drug: Intravenuse Alteplase

SUMMARY:
Ischemic stroke of the spinal cord is a rare disease accounting for about 1% of all ischemic events in the central nervous system (CNS). In most cases the consequences are catastrophic, with a high rate of severe functional disability and mortality rate up to 30%.

Ischemic stroke of the spinal cord can arise from:

1. Dissection of the aorta.
2. Aneurism in the aorta.
3. Atherosclerotic disease of the aorta or vertebral arteries.
4. Spinal surgeries.
5. Spinal AVM.
6. Embolism from cardiac origin.
7. Occlusion of radicular artery. Onset is usually sudden, reaching maximal intensity in hours until the patient becomes paralyzed in two or in all four limbs. In most cases the damage is in the Anterior Spinal Artery (ASA). The disease is expressed with motor weakness accompanied by disturbance of temperature and superficial sensation, urinary retention or bowel disorder, with preserved position and vibration sense.

The differential diagnosis of ischemic spinal cord includes diseases such as acute myelitis of the spinal cord or acute demyelinating polyneuropathy like Guillan Barree Syndrome (GBS). Therefore in order to reach the appropriate diagnosis in most cases an urgent MRI of the spinal cord is necessary upon arrival in the emergency department.

One of the treatments to acute ischemic stroke is providing thrombolysis. As tested and validated in numerous studies for ischemic events in the brain, until today no validated study in ischemic spinal stroke using thrombolysis has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with vascular risk factors
2. Patients with sudden weakness of the lower or upper limbs together with bowel disorder.
3. Window treatment - not over 6 hours since the start of the event till the start of the treatment.
4. Patient without dissection of the aorta in the abdomen.
5. Patient without contraindication to IVtPA.
6. Patient with no etiology found after clarification.

Exclusion Criteria:

1. Refusal to sign an ICF. 2. Reason for weakness is known. 3. Patient with contraindication IVtPA.

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Modified Ranking Scale (mRS) | 3 month post thrombolysis

CONTACTS AND LOCATIONS:
Overall Officials: Israel Steiner, Professor, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petach Tiqva, Central District, Israel